CLINICAL TRIAL: NCT01306981
Title: A Prospective, Randomised Controlled Trial of Ranibizumab Pre-treatment in Diabetic Vitrectomy - a Pilot Study
Brief Title: Ranibizumab in Diabetic Vitrectomy. A Prospective, Randomised Controlled Trial of Ranibizumab Pre-treatment in Diabetic Vitrectomy - a Pilot Study
Acronym: RaDiVit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAIJ1006
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Retinopathy; Retinal Neovascularisation
Keywords: Diabetes Mellitus; Diabetes Complications; Retinal Diseases; Endothelial Growth Factors; Monoclonal Antibodies; Ranibizumab; Vitrectomy; Vitreoretinal Surgery
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Neovascularization; Diabetes Mellitus; Diabetes Complications; Retinal Diseases | interventions — Ranibizumab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab (Experimental)
  Interventions: Drug: Ranibizumab
- Saline (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injection of ranibizumab, 0.5mg in 0.05ml
  Other Names: Lucentis
  Arms: Ranibizumab
Drug: Saline — Subconjunctival injection of 0.05ml saline 0.9% w/v
  Arms: Saline

SUMMARY:
This study will evaluate the effect of ranibizumab on patients undergoing vitrectomy surgery for the complications of diabetic retinopathy.

Vitrectomy surgery can be difficult and bleeding after the operation can reduce vision for patients. Our hypothesis is that injection into the eye of ranibizumab one week before surgery will make the surgery easier, reduce complications and improve outcome.

In this trial, patients will be randomly allocated to receive either ranibizumab injection or a placebo injection of saline. Neither the patient, their surgeon, nor the study investigators will know which they have received so that a fair comparison can be made.

DETAILED DESCRIPTION:
The RaDiVit study is a pilot randomised controlled trial to evaluate the effect of ranibizumab as an adjunct to diabetic vitrectomy surgery.

Patients with complications of proliferative diabetic retinopathy who require vitrectomy surgery will be recruited to this study. Baseline tests will be performed, including refracted visual acuity, B-scan ultrasound, OCT scanning, colour fundus photography and fundus fluorescein angiography. Patients will be randomised 1:1 to receive either ranibizumab intravitreal injection or saline subconjunctival injection.

One week later, surgery will be carried out. The baseline tests will be repeated on the day of surgery to examine for any discernible difference between the two groups one week after treatment. Surgery will be video recorded and detailed assessments of the operative details carried out.

A vitreous sample and a paired serum sample will be taken at the time of surgery to compare levels of ranibizumab and related cytokines.

Follow up visits will take place at six and twelve weeks. Assessments at that point will include:

* visual acuity
* OCT scan
* colour fundus photography and fundus fluorescein angiography

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex aged 18 years or over
2. Diagnosis of diabetes mellitus (type 1 or type 2). Any one of the following will be considered to be sufficient evidence that diabetes is present:

   * Current regular use of insulin for the treatment of diabetes
   * Current regular use of oral anti-hyperglycaemic agents for the treatment of diabetes
   * Documented diabetes by ADA and/or WHO criteria (see Procedures Manual for Diagnosis of Diabetes)
3. Proliferative diabetic retinopathy with complications of this requiring vitrectomy surgery with anticipated delamination of pre-retinal fibrovascular complexes
4. Ability to return for study visits
5. Ability to give informed consent throughout the duration of the study

Exclusion Criteria:

1. Hypersensitivity to the active substance or to any of the excipients.
2. Active or suspected ocular or periocular infections.
3. Vitreous haemorrhage presumed to be caused by vitreous traction on a single, focal point of vitreoretinal attachment
4. Cataract that, in the opinion of the investigators, would be significant enough to impair the view during surgery
5. Active severe intraocular inflammation
6. Previous vitrectomy surgery on study eye
7. Vision in fellow eye 3/60 or worse
8. Uncontrolled glaucoma
9. History of stroke, peripheral vascular disease, angina or myocardial infarction within six months prior to randomisation
10. Systemic anti-VEGF or pro-VEGF treatment within 3 months prior to randomisation
11. Pregnancy or lactation
12. Male or female unwilling to use contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03-30 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-03-12 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity | 12 weeks post-op

SECONDARY OUTCOMES:
Ease of performing vitrectomy surgery | One week post injection
  Assessed by surgical scoring systems and counting tool usage
Incidence of post-operative vitreous haemorrhage | 6 weeks post-op
Extent of retinal neovascularisation | 6 weeks post-op
Extent of tractional retinal detachment | 1 week post-injection
  Assessed by serial B-scan ultrasound
Extent of macular perfusion | 12 weeks post-op
  Assessed by fundus fluorescein angiography
Vitreous and serum levels of ranibizumab and related cytokines | One week post-injection
  Samples to be taken on day of surgery
Incidence of post-operative vitreous haemorrhage | 12 weeks post-op
Extent of retinal neovascularisation | 12 weeks post-op

CONTACTS AND LOCATIONS:
Overall Officials: James W Bainbridge, MA PhD FRCOphth, Principal Investigator — Moorfields Eye Hospital and UCL Institute of Ophthalmology Biomedical Research Centre for Ophthalmology
Locations (1):
- Moorfields Eye Hospital, London, United Kingdom

REFERENCES:
- [Derived] Dervenis P, Dervenis N, Smith JM, Steel DH. Anti-vascular endothelial growth factors in combination with vitrectomy for complications of proliferative diabetic retinopathy. Cochrane Database Syst Rev. 2023 May 31;5(5):CD008214. doi: 10.1002/14651858.CD008214.pub4. PMID 37260074